CLINICAL TRIAL: NCT01867944
Title: A Randomized Controlled Trial of Perineal Self-Acupressure for Chronic Constipation
Brief Title: Perineal Self-Acupressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-000738
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Constipation; Constipation; Hemorrhoids
Keywords: Chronic constipation; Hemorrhoids; Acupressure
MeSH Terms: conditions — Constipation; Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineal Self-Acupressure (Experimental): Participants in this group (intervention group) will receive education in perineal self-acupressure in addition to education in conventional treatment options for constipation.
  Interventions: Behavioral: Perineal Self-Acupressure
- Educational Control (Active Comparator): Participants in this group (the control group) will receive education in conventional treatment options for chronic constipation.
  Interventions: Behavioral: Educational Control

INTERVENTIONS:
Behavioral: Perineal Self-Acupressure — The core of the technique is to have subjects repeatedly press on and massage their perineum before defecation to fragment and soften the stool before it passes the lower rectum and anus.
  Arms: Perineal Self-Acupressure
Behavioral: Educational Control — Education on conventional treatment options for chronic constipation.
  Arms: Educational Control

SUMMARY:
The primary aim of this study is to test a non-medicinal technique for chronic constipation. The core of the technique is to have subjects repeatedly press on and massage their perineum before defecation to fragment and soften the stool before it passes the lower rectum and anus. The technique will be evaluated as a complementary treatment to standard treatment of constipation (patient educational materials about treatments such as stool softeners, laxatives fiber supplements, and increased exercise). Although this technique has been studied for other conditions (for example in pregnant women to prevent birthing-related injuries), and it is recommended anecdotally by some physicians, this would be the first time it will be studied for chronic constipation in a randomized, controlled clinical trial.

$50 dollars in compensation is provided for about an hour of participant's time.

ELIGIBILITY:
Inclusion Criteria:

* Must have experienced the following symptoms for at least three months:

  * Straining during at least 25 percent of defecations
  * Lumpy or hard stools in at least 25 percent of defecations
  * Sensation of incomplete evacuation for at least 25 percent of defecations
  * Sensation of anorectal obstruction/blockage for at least 25 percent of defecations
  * Manual maneuvers to facilitate at least 25 percent of defecations (eg, digital evacuation, support of the pelvic floor)
  * Fewer than three defecations per week
* Must have experienced one or more of those symptoms at least six months ago.

Exclusion Criteria:

* Younger than 18 years old.
* Pregnant women.
* Significant weight loss (more than 10% of usual body weight in the preceding 6 months).
* History of blood mixed in stool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Constipation Quality of Life Questionnaire | 1 month
  Constipation related health-related quality of life by means of Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL).

SECONDARY OUTCOMES:
Modified Bowel Function Index and Hemorrhoid Questionnaire | 1 month
  A modified version of the bowel function index for patient self-completion, as well as original questions to measure change in hemorrhoid impact
SF-12 | 1 month
  Questions regarding health related quality of life (HRQOL) from the Short Form (12) Health Survey version 2 questionnaire (SF-12v2).

OTHER OUTCOMES:
Technique and Educational Material Effectiveness | 1 month
  Unique questions regarding use of and effectiveness of technique and educational materials.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan B Abbott, MD, JD, MTOM, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for East-West Medicine, Los Angeles, California, United States

REFERENCES:
- [Result] Abbott R, Ayres I, Hui E, Hui KK. Effect of perineal self-acupressure on constipation: a randomized controlled trial. J Gen Intern Med. 2015 Apr;30(4):434-9. doi: 10.1007/s11606-014-3084-6. Epub 2014 Nov 18. PMID 25403522